CLINICAL TRIAL: NCT03259412
Title: Effect of Combined Fatty Acid Supplementation and Eccentric Exercise Training on Exercise Performance, Inflammation, Gene Expression and Epigenetic Signatures
Brief Title: Effect of Combined Fatty Acid Supplementation and Eccentric Exercise Training on Exercise Performance
Acronym: FAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Lynsey Wilson, Technical Tutor in Exercise Physiology/ PhD Student, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LoughboroughU
Record Dates: First submitted 2017-08-04; First posted 2017-08-23 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Exercise-induced Inflammation
MeSH Terms: interventions — Fish Oils; Fatty Acids, Omega-3; Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish Oil (Experimental): Fish oil 5.1g/ day - Premium Omega-3, Norwegian Pure-3, Oslo, Norway
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Olive Oil 6g/ day - Premium Omega-3, Norwegian Pure-3, Oslo, Norway
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish Oil Capsule
  Other Names: n-3 PUFA, Omega-3
  Arms: Fish Oil
Dietary Supplement: Placebo — Olive Oil capsule manufactured to mimic fish oil capsule
  Other Names: Olive Oil
  Arms: Placebo

SUMMARY:
The aim of the study is to determine whether fish oil (specifically omega-3 long chain polyunsaturated fatty acids [EPA-DHA]) supplementation can enhance eccentric resistance exercise performance when combined with a resistance exercise training study. The investigators aim to establish the potential mechanisms that might mediate performance changes at a cellular level.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Healthy

Exclusion Criteria:

* Resistance exercise training within the past 6 months
* Vitamin or fish oil supplementation over the past 6 months
* Habitual use of anti-inflammatory drugs
* History of heart disease
* History of coagulation/bleeding disorder
* History of metabolic disease
* Serious allergy
* Known to have blood-borne virus
* Females (Due to differences in cell membrane incorporation of Omega-3 between the sexes and the testing schedule being unable to fit in with menstrual cycle, altering the blood markers that are being measured)
* Currently no symptoms of general illness

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Strength | Change from baseline strength at 11 weeks
  Quadriceps and Hamstring strength using an isokinetic dynamometer
Leg power | Change from baseline strength at 11 weeks
  Dynamic leg power assessed through jump height on force platform

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey S Wilson, MSc, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No